CLINICAL TRIAL: NCT07161973
Title: Effect of Dietary Nitrate on Immobilization-induced Changes in Skeletal Muscle
Brief Title: Effect of Dietary Nitrate on Immobilization-induced Changes in Skeletal Muscle in Young Healthy Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Coggan, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28101
Record Dates: First submitted 2025-08-08; First posted 2025-09-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mitochondrial Energetics; Dietary Nitrate; Disuse Atrophy (Muscle) of Lower Leg
Keywords: Dietary Nitrate; Immobilization
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate (Experimental): Nitrate-rich beetroot juice
  Interventions: Dietary Supplement: Beetroot Juice - Active
- Placebo (Placebo Comparator): Nitrate-free beetroot juice
  Interventions: Dietary Supplement: Placebo Beetroot Juice Without Nitrate

INTERVENTIONS:
Dietary Supplement: Beetroot Juice - Active — Nitrate-rich beetroot juice
  Arms: Nitrate
Dietary Supplement: Placebo Beetroot Juice Without Nitrate — Nitrate-free beetroot juice
  Arms: Placebo

SUMMARY:
Diminished use of skeletal muscle, such as occurs with many chronic diseases (e.g., heart failure or cancer cachexia), denervation, bedrest, immobilization (e.g., limb casting or bracing), etc., is a common clinical condition affecting untold millions of individuals each year. Such disuse leads to a rapid decline in muscle fiber area and hence whole muscle size, contributing to a decrease in strength, speed, and power as well as alterations in energy metabolism. Collectively, these changes lead to reduced physical function and contribute to the seriousness of any disease, illness (e.g., pneumonia), surgery (e.g., joint replacement), or injury (e.g., broken bone) accompanied by decreased muscular activity. Currently, there are no effective pharmacological treatments to prevent disuse-associated muscle wasting in humans.

The above-described effects of disuse appear to be due, at least in part, to a decrease in nitric oxide (NO) bioavailability. Reduced synthesis of NO and/or increased NO destruction (due to increased production of oxygen free radicals) likely contributes to the mitochondrial changes, energetic abnormalities, and muscle atrophy resulting from immobilization. The objective of this study is to investigate the potential benefits of dietary nitrate supplementation on immobilization-induced changes in muscle contractile function and mitochondrial respiratory capacity in young healthy men. Our disuse-induced muscle atrophy model will involve wearing a knee brace for a period of 14 d.

DETAILED DESCRIPTION:
Diminished use of skeletal muscle, such as occurs with many chronic diseases (e.g., heart failure or cancer cachexia), denervation, bedrest, immobilization (e.g., limb casting or bracing), etc., is a common clinical condition aﬀecting untold millions of individuals each year. Such disuse leads to a rapid decline in muscle fiber area and hence whole muscle size, contributing to a decrease in strength, i.e., a reduction in the maximal force-generating capacity of muscle. There are also reductions in the maximal shortening velocity, and hence maximal power, of muscle, as well as alterations in energy metabolism, i.e., reduced aerobic ATP production and increased reliance on glycolysis for energy. This energetic shift likely impairs the ability of muscle to perform and recover from repeated contractions. Collectively, these changes lead to reduced physical function and contribute to increased morbidity and possibly even mortality following any disease, illness (e.g., pneumonia), surgery (e.g., joint replacement), or injury (e.g., broken bone) accompanied by decreased muscular activity. Currently, there are no eﬀective pharmacological treatments to prevent disuse-associated muscle wasting in humans.

The decline in muscle mass with disuse is due in part to downregulation of the PI3K/Akt/mTOR pathway, resulting in a reduction in the rate of protein synthesis and an increase in the rate of protein degradation, the latter due to the combined eﬀects of activation of the ubiquitin proteasome, autophagic, calpain, and caspase-3 proteolytic systems. A major factor driving these alterations in protein synthesis and degradation and hence the contractile and metabolic changes described above is a decrease in mitochondrial respiratory capacity.

Reduced mitochondrial volume, fragmentation of mitochondria resulting from disturbances in fusion/fission, increased production of reactive oxygen species (ROS), and accumulation of mitochondrial DNA (mtDNA) mutations lead to greater adenine nucleotide (ATP, ADP, and AMP) degradation, which serves to serve to activate proteolysis in part via AMPK-FoxO signaling. In support of a central role of mitochondria, overexpression of PGC1α, which induces mitochondrial biogenesis, preserves respiratory capacity and cellular energetics and minimizes atrophy resulting from denervation, hindlimb unloading, or immobilization in mouse muscle. Furthermore, administration of omega-3 fatty acids has been shown to attenuate immobilization-induced reductions in both mitochondrial bioenergetics and muscle mass in humans. The above-described eﬀects of disuse appear to be due, at least in part, to a decrease in nitric oxide (NO) bioavailability. Normal levels of NO are critical in maintaining muscle structure and function, e.g., by stimulating mitochondrial biogenesis, minimizing ROS production, suppressing calpain activation, etc. However, muscle disuse is accompanied by a decline in NO concentration, as indirectly demonstrated by a dramatic reduction in cGMP levels following denervation and directly demonstrated using electron spin resonance following spaceflight. This reduction in NO production is apparently the result of a decrease in the expression of mRNA and protein for NOS1 (nNOS), the primary isoenzyme responsible for NO production.

Dietary NO3-, a source of NO, has recently been shown to prevent immobilization-induced changes in skeletal muscle in mice. However, whether this is also true in humans is not known in muscle. Thus, reduced synthesis NO and/or increased NO destruction (due to increased ROS production) likely contribute to the mitochondrial changes, energetic abnormalities, and muscle atrophy resulting from immobilization. In support of this hypothesis, L-arginine administration has been shown to attenuate atrophy of the soleus during hindlimb suspension. Furthermore, mechanical stimulation of the plantar surface of the foot has been demonstrated to prevent or attenuate many of the changes in muscle during hindlimb immobilization in mice via an NO-dependent mechanism. Given the above, another dietary intervention with potential to mitigate disuse-induced changes in mitochondria is inorganic nitrate (NO3 -), a source of nitric oxide (NO) via the enterosalivary NO3- → nitrite (NO3-)

→ NO pathway. In both rodents and humans, dietary NO3- has been found to protect mitochondrial bioenergetics in numerous situations associated with impaired mitochondrial function, i.e., chemotherapy, high fat diet, obesity, diabetes . Furthermore, Petrick et al. recently reported that in mice NO3- intake prevented changes in mitochondrial respiration and ROS production due to hindlimb immobilization. This treatment, however, did not alter the extent of atrophy, nor were Petrick et al. able to determine the mechanism by which dietary NO3- maintained mitochondrial function. Nonetheless, these intriguing preclinical findings suggest that NO3- supplementation may ameliorate at least some of the negative consequences of muscle disuse in humans.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18-44
* Above the minimum threshold of the IPAQ questionnaire
* Below the maximum threshold of the IPAQ questionnaire

Exclusion Criteria:

* Men and women <18 or >44 years of age
* Unable to provide informed consent
* Known clotting disorder
* Previous history of deep vein thrombosis
* Injury to either leg resulting in reduced mobility in the previous year
* Currently dieting or weight instability for the past 3 months
* Epileptic
* Pacemaker or other implantable heart device
* Currently taking antibiotics
* Current smoker
* Stage II hypertension (resting blood pressure >140/>90)
* Previously undergone a revascularization procedure involving a vascular graft or stenting of the femoral or popliteal arteries
* Those taking phosphodiesterase inhibitors (e.g., Viagra), proton pump inhibitors, antacids, xanthine oxidase inhibitors, hormonal contraceptives or on hormone replacement therapy
* An answer of yes to any of the seven questions on the first page of the Physical Activity Readiness Questionnaire (PAR-Q. These exclusions include the following:

  * If participant's doctor has ever said that he/she has a heart condition and that he/she should only do physical activity recommended by a doctor
  * Pain in chest when doing physical activity
  * In past month, chest pain when not doing physical activity
  * If participant has ever lost balance because of dizziness or has ever lost consciousness
  * Muscle, bone, or joint problem that could be made worse by physical activity
  * Currently on prescribed drugs for blood pressure or heart condition.
  * If the participant knows of any other reason he/she should not do physical activity.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mitochondrial function | 14 days
  Muscle mitochondrial respiratory capacity assessed in vitro using high resolution respirometry and in vivo using a near infrared spectroscopy/occlusion protocol

SECONDARY OUTCOMES:
Muscle strength | 14 days
  Muscle strength as assess using isokinetic dynamometry
Muscle speed | 14 days
  Muscle speed as assess using isokinetic dynamometry
Muscle power | 14 days
  Muscle power as assessed using isokinetic dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Coggan, PhD, Principal Investigator — Indiana University Indianapolis
Locations (1):
- Indiana University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-PHI individual participant data will be shared upon reasonable request.
Time Frame: Data will be made available upon completion of the study and publication of the final results.